CLINICAL TRIAL: NCT04206475
Title: Feasibility Randomized Trial for an Intensive Memory-Focused Training Program for School Aged Children With Acquired Brain Injury.
Brief Title: Feasibility Randomized Trial for an Intensive Memory-Focused Training Program for School Aged Children With Acquired br.Inj.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Id. No.08/19_Oss
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: an intensive program specific to the training and re-adaptation of memory function in children versus standard rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IM-FTP (Experimental): rehabilitated over 1-month through IM-FTP, including physio-kinesis/occupational, speech, and neuropsychology treatments
  Interventions: Other: rehabilitation; Other: Intensive Memory-Focused Training Program (IM-FTP)
- standard rehabilitation (Active Comparator): physio-kinesis, occupational, speech, and neuropsychology treatments
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — the rehabilitation program consisted of an intensive treatment lasting 4 weeks, and including 3 daily interventions each working day (5 working days per week, for a total of 20 days of treatment and 60 sessions). The 3 daily sessions were organized as follows:
  1 physio-kinesis and/or occupational therapy, 1 speech therapy, and 1 neuro-psychology treatment.
  Each session lasted 45 minutes.
Other: Intensive Memory-Focused Training Program (IM-FTP) — During each session, the patient was engaged in a one-to-one interaction with the therapist. Overall, the treatment targeted the following memory subfunctions: verbal and visuo-spatial short-term memory, verbal and visuo-spatial long-term memory, working memory and procedural memory
  Arms: IM-FTP

SUMMARY:
Memory deficits are common sequelae of pediatric Acquired Brain Injury (ABI). Only methods for non-focused cognitive remediation are available to the pediatric field. The aims of this feasibility trial are the description, implementation, and test of an intensive program specific to the training and re-adaptation of memory function in children (IM-FTP). Method: Eleven children and adolescents with ABI (mean age at injury=12.2 years, brain tumor survivors excluded) were clinically assessed and rehabilitated over 1-month through IM-FTP, including physio-kinesis/occupational, speech, and neuropsychology treatments. Each patient received a psychometric evaluation and a brain functional MRI at enrollment and at discharge. Ten pediatric controls with ABI (mean age at injury=13.8 years) were clinically assessed, and rehabilitated through a standard program.

ELIGIBILITY:
Inclusion Criteria:

* i) age at first assessment between 6 and 18 years;
* ii) time between injury and first assessment <3 months;
* iii) documented evidence of a severe ABI of traumatic or non-traumatic (i.e. anoxic, vascular or infectious) etiology, as indicated by a Glasgow Coma Scale (GCS, [26]), score ≤8 at insult;
* iv) presence of severe memory impairment, as assessed at first evaluation;
* v) sufficient attentive skills for attending a simple task and understanding simple commands/directions, and sufficient verbal comprehension for executing simple procedures/exercises;
* vi) absence of congenital pathology or disability previous to the injury;
* vii) medical records sufficiently detailed to determine the injury severity and neurological findings;
* viii) absence of severe motor or sensitive deficits.

Exclusion Criteria:

* none

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-02-03 (Actual)

PRIMARY OUTCOMES:
Psychometric evaluation | 4 weeks
  At both time points, the patients were administered the Rey- Osterrieth complex figure test (REY), the test for immediate and delayed memory of a list of words of the Italian 'Batteria di Valutazione Neuropsicologica' (BVN) battery (BVNLi and BVNLd, respectively), the test for immediate and delayed recall in prose memory of the Italian BVN battery (BVNPi and BVNPd), the test for immediate and delayed recall in positional memory supra-span (SUPRASPANi and SUPRASPANd), and the Italian TEMA test for the learning of couples of related and unrelated words (TEMA)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No